CLINICAL TRIAL: NCT05356234
Title: Randomized Controlled Trial of the Jewish Family and Children's Service of the Suncoast, Inc.
Brief Title: Ignite Study of the Jewish Family and Children's Service of the Suncoast, Inc.
Acronym: Ignite
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish Family & Children's Service of the Suncoast, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20220421
Record Dates: First submitted 2022-04-22; First posted 2022-05-02 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Intervention; Wait-List Control
Keywords: Healthy parent and child relationships; Economic self-sufficiency
MeSH Terms: interventions — Association

STUDY DESIGN:
Intervention Model Description: The Intervention group will start with assigning a Case Manager and conducting a series of workshops addressing responsible parenting and marriage and relationships as well as a complement of employment services and comprehensive case management.
Who Masked: Outcomes Assessor
Masking Description: The outside evaluators will remain blind to each condition throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Intervention: Responsible Parenting, Relationships, and Employment Services (Experimental): Experimental: A series of workshops addressing responsible parenting and marriage and relationships as well as a complement of employment services and comprehensive case management will be conducted over a 12-week period.
  Interventions: Behavioral: Treatment Intervention: Responsible Parenting, Relationships, and Employment Services
- Wait-List Control (No Intervention): The Wait-List Control group will be placed on a wait-list and offered services as soon as they complete the study's final 24-week follow-up measures. Wait-List Control participants will not be assigned a Case Manager and will not receive any comparable services from our agency until they complete their 24-week measures.

INTERVENTIONS:
Behavioral: Treatment Intervention: Responsible Parenting, Relationships, and Employment Services — The Intervention group will be assigned a Case Manager and placed in the next available On My Shoulders (OMS) curriculum that offers strategies to help individuals develop a strong and healthy self in the service of making current and/or future relationships of all forms (parent-child, romantic, family, work) successful and satisfying. This curriculum is intended to equip men (and, where applicable, women) with the skills they need to build and nurture healthy relationships. This curriculum should help participants improve family functioning. Additionally, Transforming Impossible into Possible (TIP) financial literacy curriculum will be utilized to help participants increase job retention for those currently employed, improve wages through additional educational and training opportunities, and learn skills to better manage family finances. This curriculum should help participants increase economic stability and mobility.
  Arms: Treatment Intervention: Responsible Parenting, Relationships, and Employment Services

SUMMARY:
The goals of the program are to help struggling fathers and father figures improve the parent-child relationship, sustain healthy marriages and relationships (and help those who are single identify ways to enter into safe and supportive relationships that may ultimately lead to marriage), and identify and support fathers in their economic stability and employment objectives. These outcomes will be achieved through a series of workshops addressing responsible parenting and marriage and relationships as well as a complement of employment services and comprehensive case management. Additional services needed by participants will be identified and provided either through wraparound programming provided by JFCS or through collaborative agreements with local partner agencies. Additionally, Ignite will incorporate a comprehensive employment program combining both job and career advancement.

DETAILED DESCRIPTION:
In each full year of the grant, this program will serve a minimum of 250 community-based fathers or expectant fathers (custodial or noncustodial) who are age 18 and older and who have a child or children under the age of 24. While the program will be targeted to fathers, mothers may also be served, as might individuals who play a father figure role such as adoptive fathers, foster fathers, grandfathers, etc. Ignite will serve the geographic area of Sarasota, Manatee, and Charlotte counties on the Gulf Coast of Florida. The goals of the program are to help struggling fathers and father figures improve the parent-child relationship, sustain healthy marriages and relationships (and help those who are single identify ways to enter into safe and supportive relationships that may ultimately lead to marriage), and identify and support fathers in their economic stability and employment objectives. These outcomes will be achieved through the provision of a series of workshops addressing responsible parenting and marriage and relationships as well as a complement of employment services and comprehensive case management. Additional services needed by participants will be identified and provided either through the extensive wraparound programming provided by JFCS or through collaborative agreements with local partner agencies.

Additionally, Ignite will incorporate a comprehensive employment program combining both job and career advancement. This will help fathers in crisis reach improved financial stability, which will in turn improve the ability of individual participants to be better parents and better partners, furthering the goals to foster more stable parent-child relationships and promote healthy marriages in the region. Nationwide 35% of children live in single parent families. Growing up in a single-parent family increases a child's risk of growing up poor, becoming a teen parent, dropping out of school, and disconnecting from the labor market. Coupled with its successful history of providing healthy marriage programming, JFCS as an agency is well-positioned to help families in crisis (both due to current economic conditions and in more long-term tenuous situations) become more stable and self-sufficient. Notable within our local demographic data is a significantly higher than average rate of unemployment and higher percentages of income in the past 30 days less than $500. Understanding the inextricable link between financial security and family stability, Ignite is truly targeting and reaching the most vulnerable individuals based solely on economic risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 or older
2. Have a child or children under the age of 24
3. Interested in improving the parent-child relationship, sustain healthy marriages and relationships, and economic stability and employment objectives
4. Resides in Sarasota, Manatee, and Charlotte counties on the Gulf Coast of Florida

Exclusion Criteria:

1. Under age 18
2. Does not reside in Sarasota, Manatee, and Charlotte counties on the Gulf Coast of Florida

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 675 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Family Environment Survey (FES) | 24 weeks
  The FES was developed to measure social and environmental characteristics of families. Face and content validity are supported by clear statements about family situations that relate to subscale domains, and the measure can differentiate between distressed and normal family samples.
Revised Dyadic Adjustment Scale (RDAS) | 24 weeks
  The RDAS is a 32-item self-report standardized measure with 4 subscales: (1) Dyadic Consensus, (2) Dyadic Satisfaction, (3) Affectional Expression, and (4) Dyadic Cohesion as well as a total score.
Perceived Employment Barriers Scale (PEBS) | 24 weeks
  The PEBS is a 20-item scale developed to measure barriers to employment including the following subscales: (1) Physical and mental health, (2) Labor market exclusion, (3) Child care, (4) Human capital, and (5) Soft skills. The measure is a Likert-type scale ranging from 1 to 5 where 1 indicates 'not a barrier' and 5 indicates 'strong barrier'.
Employment Hope Scale (EHS) | 24 weeks
  The EHS is a 14-item scale developed to measure psychological self-sufficiency with two subscales: (1) psychological empowerment, and (2) goal-oriented pathways. This is a Likert-type scale ranging from 0 to 10 where 0 indicates 'strongly disagree' and 10 indicates 'strongly agree'.

CONTACTS AND LOCATIONS:
Overall Officials: Katelyn Kopakin, MA, Study Director — Jewish Family Children's Services of the Suncoast, Inc.
Locations (1):
- Jewish Family and Children Service of the Suncoast, Inc., Sarasota, Florida, United States